CLINICAL TRIAL: NCT06562712
Title: Evaluation of Bilateral Internal Iliac Artery Balloon Occlusion in Placenta Accreta Spectrum Management: A Randomized Controlled Trial
Brief Title: Evaluation of Bilateral Internal Iliac Artery Balloon Occlusion in Placenta Accreta Spectrum Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed Ibrahim Adel Eleissawy, Lecturer of Vascular and Endovascular Surgery, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 36264PR753/7/24
Record Dates: First submitted 2024-08-15; First posted 2024-08-20 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Internal Iliac Artery; Balloon Occlusion; Placenta Accreta Spectrum
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional management (Active Comparator): Patients will be subjected to conventional management for placenta accreta spectrum.
  Interventions: Procedure: Conventional management
- Bilateral internal iliac artery balloon occlusion (Experimental): Patients will be subjected to bilateral internal iliac artery balloon occlusion for placenta accreta spectrum.
  Interventions: Procedure: Bilateral internal iliac artery balloon occlusion

INTERVENTIONS:
Procedure: Conventional management — Patients will be subjected to conventional management for placenta accreta spectrum.
  Arms: Conventional management
Procedure: Bilateral internal iliac artery balloon occlusion — Patients will be subjected to bilateral internal iliac artery balloon occlusion for placenta accreta spectrum.
  Arms: Bilateral internal iliac artery balloon occlusion

SUMMARY:
This study aims to evaluate the efficacy and safety of bilateral internal iliac artery balloon occlusion in the management of the placenta accreta spectrum.

DETAILED DESCRIPTION:
Placenta accreta spectrum (PAS) is abnormal placental adhesion beyond superficial myometrium, which includes placenta accreta, placenta increta, and placenta percreta.

However, there is a desire to preserve the uterus and fertility, so alternatives to hysterectomy are needed. Presently, attempts to avoid hysterectomy include reducing intraoperative hemorrhage such as uterine compression sutures, intrauterine balloon tamponade, pelvic artery ligation, and spiral suturing of the lower uterine segment. Intrauterine balloon tamponade may increase CS scar dehiscence, uterine rupture, and infection. Combined with compression sutures, it may induce uterine necrosis.

Placement of balloons in the bilateral internal iliac arteries before caesarean section can reduce uterine artery pressure and intraoperative blood loss during balloon inflation, thus temporarily blocking the main blood supply of the uterus, helping to expose the visual field, shortening the operation time during surgery, and leading to opportunities for timely adjustments to the operative plan during surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 40 years.
* Women with placenta accreta spectrum based on ultrasound (US) and/or magnetic resonance imaging (MRI) findings.

Exclusion Criteria:

* Women with a bleeding disorder.
* History of known allergy to contrast media.
* Women with Impaired renal function.
* Emergency cesarean section.
* Women had severe attack of bleeding before the operation affecting patient's general condition.
* Women had previous four or more cesarean scars.
* If ultrasound (US) and magnetic resonance imaging (MRI) suspect the presence of placenta accrete preoperative, then intraoperative the placenta is found to have normal adhesion to the uterine wall, this case will be excluded.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women with placenta accreta spectrum
Enrollment: 30 (Actual)
Dates: Start 2024-08-20 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Amount of intraoperative blood loss | Intraoperatively
  The amount of intraoperative blood loss will be calculated with reference to the contents of the suction apparatus and to weight of the surgical pads and the hemoglobin concentration difference, immediate preoperative (the morning of cesarean delivery) and postoperative (immediately after cesarean delivery) hemoglobin levels.

SECONDARY OUTCOMES:
Operation time | From the start till the end of surgery
  Operation time will be recorded from start till end of surgery.
Number of blood products units transfused | 24 hours postoperatively
  Number of blood products units transfused will be recorded.
Hospitalization length | 28 days postoperatively
  Hospitalization length will be recorded from admission till discharge from hospital.
Incidence of hysterectomy | 24 hours postoperatively
  Incidence of hysterectomy will be recorded.
Intensive Care Unit (ICU) admission rate | 24 hours postoperatively
  Intensive Care Unit (ICU) admission rate will be recorded.
Intraoperative complications | Intraoperatively
  Intraoperative complications such as bladder injury, ureteric ligature, and uterine atony will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.